CLINICAL TRIAL: NCT03908918
Title: Mind and Body: A Clinical Trial Evaluation of a Smartphone App-based Mindfulness Intervention to Support Psychosocial Resilience in Aging Patients
Brief Title: Mind and Body:A Clinical Trial Evaluation of a Smartphone App-based Mindfulness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Providence Healthcare (Other)
Responsible Party: Principal Investigator, Rachel Devitt, Professional Practice Leader, Occupational Therapy and Manager, Clinical Research at Providence Healthcare, Providence Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 123
Record Dates: First submitted 2019-03-19; First posted 2019-04-09 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Psychological Stress; Psychological Distress; Rehabilitation
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Mobile-app delivered mindfulness intervention. Dosage: 4 times per week for 4 weeks
  Interventions: Other: Mindfulness app
- Waitlist control (Other): Waitlist control - receiving the app after 6 months
  Interventions: Other: Mindfulness app

INTERVENTIONS:
Other: Mindfulness app — Mobile app-delivered mindfulness intervention delivered over 4 weeks.
  Other Names: Am

SUMMARY:
This study evaluates the use of a mobile-app delivered mindfulness-based intervention for supporting psychosocial resilience in aging patients undergoing rehabilitation treatment. Half of the patients will receive the mobile-app, while the other half will receive the app 6 months later.

DETAILED DESCRIPTION:
Although, several mobile-app based MBTs are available in the marketplace, there is scant evidence of high scientific rigor to support their therapeutic efficacy. Furthermore, the tracking of wellness outcomes, stress resilience and functioning as a result of use of a therapeutic digital product is a challenging task requiring expertise in technology. In this study, the investigators aim to investigate not only the effectiveness of an app-based MBT in aging adults, but also the mechanisms of efficacy - i.e. the therapeutic effects - of app usage, including changes in, depression, anxiety, or mood and the acceptance of the app in older adult populations. The investigators also aim to measure the Return On Investment (ROI) of mobile mindfulness on health services utilization.

The study is a randomized controlled design with 1:1 equal allocation to treatment (Experimental Am app group) or control (treatment as usual). The investigators will recruit 82 participants in total.

The Experimental group will start the 4 week Am app intervention immediately after randomization and baseline intervention questionnaires, while the wait-list control group will receive treatment as usual. Assessments are conducted at four time point: At Baseline (#1), Post-Intervention (#2), Follow-up at 3 months post baseline (#3) and Follow-up at 6 months post baseline (#4).

The clinical champions that referred the patient to the study will complete brief surveys about the quality of their appointments with the patient at two time points: At baseline (#1) and Post-Intervention (#2).

The waitlist control group will be granted access to the mindfulness intervention at 6 months post baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over the age of 40.
2. Admitted as In-Patients.
3. Access to a smart phone with data connection.
4. Willing to give time for mindfulness practice.
5. Sufficient ability to speak and read English.
6. Willingness to be randomized into immediate or waitlist groups and complete all assessments.

Exclusion Criteria:

1. Any cognitive or mental impairment that would interfere with completing questionnaires or the intervention (<6 on the Brief Screen for Cognitive Impairment) .
2. Admitted to Providence as an in-patient to long-term care or palliative care.
3. An existing smartphone app-based mindfulness practice consisting of one or more sessions per week.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Outcome: Cost of treatment; Measure: Duration of stay | 6 months
  To evaluate the cost-benefit measures of the Am smartphone-app by measuring length of stay in hospital and levels of health services utilization
  As no Electronic Health Records (EHR) are kept by Providence, a chart review, including progress notes, will be required to assess the following:
  * Date of admission.
  * Date of discharge.
Outcome: Health services utilization; measure: survey questions | 6 months
  Cost of Treatment will also be measured using patient self-reports of health services utilization at 3 and 6 months post intervention. Participants will answer five questions related to their use of health services utilization drawn from peer-reviewed literature (Van den Brink et al., 2005).
  1. Compared to the 3 months prior to the study, in the past 3 months my use of health care services has: (1) greatly decreased (2) stayed the same (3) greatly increased
  2. How many times did you visit your doctor's office visits in the last 3 months?
  3. How many times a caregiver visit you in your home in the last 3 months?
  4. How many times were you admitted to a hospital in the last 3 months.
Outcome: Cost of treatment; Measure: Discharge destination | 6 months
  Indicates whether the patient returns home, or is discharged to another care facility (e.g., long term or palliative care).
Outcome: Cost of treatment; Measure: Alternate Level of Care (ALC) assignment. | 6 months
  If Alternate Level of Care (ALC) assigned, the reasons underlying the decision. The term ALC is a clinical designation that identifies patients who no longer require the intensity of resources or services provided in their current settings and who are wait
Outcome: Cost of treatment; Measure: National Rehabilitation Reporting System (NRS) assessments. | 6 months
  The NRS minimum data set contains clinical data on functional status based on the 18-item Functional Independence Measure (FIM®) instrument.
  FIM™ is comprised of 18 items, grouped into 2 subscales - motor and cognition.
  Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.
  1. - Total assistance with helper
  2. - Maximal assistance with helper
  3. - Moderate assistance with helper
  4. - Minimal assistance with helper
  5. - Supervision or setup with helper
  6. - Modified independence with no helper
  7. - Complete independence with no helper
Outcome: Cost of treatment; Measure: Rehabilitation Patient Group (RPG) | 6 months
  The NRS gives an RPG score used to categorize patient data based on their primary reason for receiving inpatient rehabilitation services.
  Based on a patient's primary reason for receiving inpatient rehabilitation services, and using client age at admission and motor and cognitive functional status, patient's are assigned to one of 83 RPGs.
Outcome: Cost of treatment; Measure: number of clinic visits | 6 months
  Post six-month retrospective report of patients' clinic visits.

SECONDARY OUTCOMES:
Outcome: stress; Measure: NIH Toolbox Perceived Stress Fixed Form (Age 18+ v2.0) | 6 months
  To evaluate the efficacy of the Am smartphone-app to relieve symptoms of stress
  The NIH Toolbox Perceived Stress Fixed Form contains measures in the domains of emotional health and was designed for use in epidemiological and clinical trials health-related research. It was selected for inclusion and subsequent national norming for the NIH Toolbox based on its psychometric performance.
Outcome: Impact on health-related quality of life; Measure: PROMIS57 | 6 months
  To evaluate the efficacy of the Am smartphone-app for treating symptoms of anxiety, sleep disturbance, mood disturbance, and overall quality of life
  PROMIS57 is a collection of short forms containing a fixed number of items from seven PROMIS domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities). There are 8 questions per domain, and an additional pain intensity 0-10 numeric rating scale (NRS). The Profiles are universal rather than disease-specific.
Outcome: clinician reported quality of patient appointment time; measure: purpose designed survey questions | 1 month
  Survey 1
  1. How has this patient's mental health impacted the quality of time spent during your appointments with them to-date?
  2. Have you had to make last minute changes to your care plan for this patient depending on their mental state when they have come to attend appointments?
  Survey 2
  1. How has the quality of time spent during your appointments with this patient has changed over the last 4 weeks?
  2. Over the last 4 weeks, how has this patient's mental health impacted the quality of time spent during your appointments with them?
  3. Over the last 4 weeks, have you had to make last minute changes to your care plan for this patient depending on their mental state when they have come to attend appointments?
Outcome: Mood; Measure: The Am app's mood measure | 6 months
  Am quantifies the efficacy of mindfulness training on each individual user through self-reports.
  Self-reported mood will be collected by the participant's selection of mood words from Mobio's circumplex model of affect (based on Posner, Russell & Peterson, 2005). This model holds that all emotions derive from two underlying, orthogonal dimensions of emotional experience: valence and arousal. These orthogonal dimensions divide the circumplex into four quarters: low arousal - low affect; low arousal - high affect; high arousal - low affect; high arousal - high affect.
Outcome: Psychological flexibility; Measure: The Acceptance & Action Questionnaire-II | 6 months
  The Acceptance & Action Questionnaire-II (AAQ-II) was developed in order to measure psychological flexibility, and scores have been found to predict many outcomes, including mental health and work absence rates.
  The AAQ-II is a seven item, one factor measure of psychological inflexibility or experiential avoidance. The scale is scored by summing the responses. Higher scores equal greater levels of psychological inflexibility.
Outcome: User engagement; Measure: The Am app's user analytics - meditation choice and frequency | 6 months
  The time, date and type of meditation users choose while participating in the study.
Outcome: Mood, stress and heart rate; Measure: The Am app's biometric measures (Heart Rate) | 6 months
  Am quantifies the efficacy of mindfulness training on each individual user through heart rate, an objective assessment of stress made possible through computer vision (biometrics) with the mobile device camera.
Outcome: Mood, stress and heart rate; Measure: The Am app's biometric measures (respiratory rate) | 6 months
  Am quantifies the efficacy of mindfulness training on each individual user through respiratory rate, an objective assessment of stress made possible through computer vision (biometrics) with the mobile device camera.
Outcome: Mood, stress and heart rate; Measure: The Am app's biometric measures (relative blood oxygen saturation) | 6 months
  Am quantifies the efficacy of mindfulness training on each individual user through relative blood oxygen saturation, an objective assessment of stress made possible through computer vision (biometrics) with the mobile device camera.
Outcome: Stress; Measure: The Am app's stress measure | 6 months
  Am quantifies the efficacy of mindfulness training on each individual user through self-reports.
  Self-reported stress will be indicated by the participant's adjustment of a dynamic slider between the minimum score "no stress" and the maximum score "max stress" will be collected.
Outcome: Stress; Measure: The Am app's intent for practicing mindfulness measure | 6 months
  This will be based on the participants' indication as per their selection of between 1 and 3 "intent words". There are 24 options from which the participant can choose. These are divided into 6 outward intentions, and 18 inward intentions.
Outcome: User engagement; Measure: The Am app's points structure | 6 months
  Users are rewarded with in-app points according to a point structure that encourages engagement with the app.
  3. Page/screen views and dwell time.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Devitt, Principal Investigator — Providence Healthcare
Locations (1):
- Providence Healthcare, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sachs-Ericsson N, Van Orden K, Zarit S. Suicide and aging: special issue of Aging & Mental Health. Aging Ment Health. 2016;20(2):110-2. doi: 10.1080/13607863.2015.1099037. Epub 2015 Nov 7. No abstract available. PMID 26548754
- [Background] Schulze T, Maercker A, Horn AB. Mental health and multimorbidity: psychosocial adjustment as an important process for quality of life. Gerontology. 2014;60(3):249-54. doi: 10.1159/000358559. Epub 2014 Feb 28. PMID 24603025
- [Background] Rao KS, Chakraharti SK, Dongare VS, Chetana K, Ramirez CM, Koka PS, Deb KD. Antiaging Effects of an Intensive Mind and Body Therapeutic Program through Enhancement of Telomerase Activity and Adult Stem Cell Counts. J Stem Cells. 2015;10(2):107-25. PMID 27125139
- [Background] Scult M, Haime V, Jacquart J, Takahashi J, Moscowitz B, Webster A, Denninger JW, Mehta DH. A healthy aging program for older adults: effects on self-efficacy and morale. Adv Mind Body Med. 2015 Winter;29(1):26-33. PMID 25607120
- [Background] de Frias CM, Whyne E. Stress on health-related quality of life in older adults: the protective nature of mindfulness. Aging Ment Health. 2015;19(3):201-6. doi: 10.1080/13607863.2014.924090. Epub 2014 Jun 18. PMID 24940847
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Charness N, Best R, Evans J. Supportive home health care technology for older adults: Attitudes and implementation. Gerontechnology. 2016 Feb 23;15(4):233-242. doi: 10.4017/gt.2016.15.4.006.00. PMID 29033700
- [Background] Deng Z, Mo X, Liu S. Comparison of the middle-aged and older users' adoption of mobile health services in China. Int J Med Inform. 2014 Mar;83(3):210-24. doi: 10.1016/j.ijmedinf.2013.12.002. Epub 2013 Dec 16. PMID 24388129
- [Background] Nguyen T, Irizarry C, Garrett R, Downing A. Access to mobile communications by older people. Australas J Ageing. 2015 Jun;34(2):E7-E12. doi: 10.1111/ajag.12149. Epub 2014 Apr 17. PMID 24750499
- [Background] Walsh KM, Saab BJ, Farb NA. Effects of a Mindfulness Meditation App on Subjective Well-Being: Active Randomized Controlled Trial and Experience Sampling Study. JMIR Ment Health. 2019 Jan 8;6(1):e10844. doi: 10.2196/10844. PMID 30622094
- [Background] Hill J, McVay JM, Walter-Ginzburg A, Mills CS, Lewis J, Lewis BE, Fillit H. Validation of a brief screen for cognitive impairment (BSCI) administered by telephone for use in the medicare population. Dis Manag. 2005 Aug;8(4):223-34. doi: 10.1089/dis.2005.8.223. PMID 16117717
- [Background] van den Brink M, van den Hout WB, Stiggelbout AM, Putter H, van de Velde CJ, Kievit J. Self-reports of health-care utilization: diary or questionnaire? Int J Technol Assess Health Care. 2005 Summer;21(3):298-304. doi: 10.1017/s0266462305050397. PMID 16110708